CLINICAL TRIAL: NCT01218204
Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Administering Multiple Oral Doses of GSK1292263 Alone and With Atorvastatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 113779
Record Dates: First submitted 2010-09-23; First posted 2010-10-11 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Dyslipidaemias; Dyslipidemias
Keywords: Pharmacodynamics; Lipids; Dyslipidemia; Safety; GSK1292263; Ezetimibe; Statin; Pharmacokinetics; Tolerability; Atorvastatin
MeSH Terms: conditions — Dyslipidemias | interventions — Atorvastatin; (1-(3-isopropyl-1,2,4-oxadiazol-5-yl)piperidin-4-yl)methyl methanesulfonate; Ezetimibe; WASH protein, Drosophila

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (16):
- Part A Run-in (Other): Subjects on stable 40mg atorvastatin > 4 weeks may raise their dose to 80mg for 2 weeks in order to qualify for Part A.
  Interventions: Drug: 80mg atorvastatin
- Part A Co-Dosing 800mg GSK1292263 (Experimental): Dosing for 14 days
  Interventions: Drug: 800mg GSK1292263
- Part B Washout (Other): Washout for 4 weeks
  Interventions: Other: Washout
- Part B Run-in 10mg atorvastatin (Active Comparator): Dosing for 4 weeks
  Interventions: Drug: 10mg atorvastatin
- Part B Run-in 80mg atorvastatin (Active Comparator): Dosing for 4 weeks
  Interventions: Drug: 80mg atorvastatin
- Part B Co-Dosing 10mg atorvastatin + 100mg GSK1292263 (Experimental): Dosing for 14 days
  Interventions: Drug: 10mg atorvastatin
- Part B Co-Dosing 10mg atorvastatin + 300mg GSK1292263 (Experimental): Dosing for 14 days
  Interventions: Drug: 300mg GSK1292263
- Part B Co-Dosing 10mg atorvastatin + 800mg GSK1292263 (Experimental): Dosing for 14 days
  Interventions: Drug: 10mg atorvastatin; Drug: 800mg GSK1292263
- Part B Co-Dosing 10mg atorvastatin + 10mg ezetimibe (Experimental): Dosing for 14 days
  Interventions: Drug: 10mg atorvastatin; Drug: 10mg ezetimibe
- Part B Dosing 100mg GSK1292263 (Experimental): Dosing for 14 days
  Interventions: Drug: 100mg GSK1292263
- Part B Dosing 300mg GSK1292263 (Experimental): Dosing for 14 days
  Interventions: Drug: 300mg GSK1292263
- Part B Dosing 800mg GSK1292263 (Experimental): Dosing for 14 days
  Interventions: Drug: 800mg GSK1292263
- Part B Dosing Placebo GSK1292263 (Experimental): Dosing for 14 days
  Interventions: Drug: GSK1292263 Placebo
- Part B Co-Dosing 80mg atorvastatin + 800mg GSK1292263 (Experimental): Dosing for 14 days
  Interventions: Drug: 80mg atorvastatin
- Part B Co-dosing 80mg atorvastatin + Placebo (GSK1292263) (Experimental): Dosing for 14 days
  Interventions: Drug: GSK1292263 Placebo
- Part B Co-Dosing 10mg atorvastatin + Placebo (GSK1292263) (Experimental): Dosing for 14 days
  Interventions: Drug: 10mg atorvastatin

INTERVENTIONS:
Drug: 10mg atorvastatin — 10mg
  Other Names: Lipitor
  Arms: Part B Co-Dosing 10mg atorvastatin + 100mg GSK1292263; Part B Co-Dosing 10mg atorvastatin + 10mg ezetimibe; Part B Co-Dosing 10mg atorvastatin + 800mg GSK1292263; Part B Co-Dosing 10mg atorvastatin + Placebo (GSK1292263); Part B Run-in 10mg atorvastatin
Drug: 80mg atorvastatin — 80mg
  Other Names: Lipitor
  Arms: Part A Run-in; Part B Co-Dosing 80mg atorvastatin + 800mg GSK1292263; Part B Run-in 80mg atorvastatin
Drug: GSK1292263 Placebo — Placebo
  Arms: Part B Co-dosing 80mg atorvastatin + Placebo (GSK1292263); Part B Dosing Placebo GSK1292263
Drug: 100mg GSK1292263 — 100mg
  Arms: Part B Dosing 100mg GSK1292263
Drug: 300mg GSK1292263 — 300mg
  Arms: Part B Co-Dosing 10mg atorvastatin + 300mg GSK1292263; Part B Dosing 300mg GSK1292263
Drug: 800mg GSK1292263 — 800mg
  Arms: Part A Co-Dosing 800mg GSK1292263; Part B Co-Dosing 10mg atorvastatin + 800mg GSK1292263; Part B Dosing 800mg GSK1292263
Drug: 10mg ezetimibe — 10mg
  Other Names: Zetia
  Arms: Part B Co-Dosing 10mg atorvastatin + 10mg ezetimibe
Other: Washout — No interventions - washout period
  Arms: Part B Washout

SUMMARY:
This study investigates the safety, pharmacokinetics and effects of GSK1292263 when taken alone or when co-dosed with atorvastatin to subjects with dyslipidemia.

DETAILED DESCRIPTION:
This compound has been studied in healthy subjects and subjects with type II diabetes and is now being studied in subjects with dyslipidemia. Because many patients with dyslipidemia are on statins, it is important to study how GSK1292263 behaves when taken with a potent statin, atorvastatin. The cholesterol lowering drug, ezetimibe, is included for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females of non-child-bearing-potential, aged 18-75 years who is capable of giving informed consent.
* A female subject is eligible to participate if she is of:

  * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. In questionable cases, a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol <40 pg/ml (<140 pmol/L) is confirmatory in the absence of a clear post-menopausal history.
  * Females on hormone replacement therapy (HRT) must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study.
* Male subjects must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until seven days following the last dose.
* Body weight > 50 kg (110 pounds) and body mass index (BMI) between 19.0 and 39.0 (inclusive).
* Part A: (i) Subjects who are on 80mg or 40mg atorvastatin for >= 4 weeks and are tolerating the drug well, or (ii) Subjects not on lipid-modifying therapy who have a fasting low density lipoprotein cholesterol (LDLc) >= 130mg/dL.
* In Part B at Screening: Subjects who are on statins or Vytorin treatment for >= 4 weeks.
* Part B at the end of the 4 week washout: Subjects who have a fasting LDL cholesterol of >=120mg/dL and <=180mg/dL and fasting triglycerides of >=100mg/dL and <=400mg/dL.
* Part B at the end of the 4 week run-in on atorvastatin: Subjects who are tolerating well atorvastatin 10mg or 80mg (as determined by the Investigator).
* Part B: Subjects must be willing to discontinue statins or Vytorin for the duration of the study.
* Liver enzymes, AST and ALT < 2x upper limit of normal (ULN); alkaline phosphatase and bilirubin =< 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). Subjects with Gilbert's syndrome are allowed to participate in the study.
* Average QTcB or QTcF < 450msec; or QTc < 480msec in subjects with right bundle branch block.

Exclusion Criteria:

* A medical history of the following:

  * Clinical or angiographic cardiovascular disease, including history or current evidence of coronary heart disease, heart failure, cerebrovascular disease (including stroke and transient ischemic attack [mini-stroke]), peripheral vascular disease. Subjects pending diagnostic procedures for any of those conditions at the time of screening will not be eligible for participation.
  * Homozygous familial hypercholesterolemia or family history of familial hypercholesterolemia (Part B only). Note: Subjects with heterozygous familial hypercholesterolemia on 80mg atorvastatin who are tolerating this drug well and fulfill the other eligibility criteria may participate in Part A only.
  * History of recurrent or unexplained muscle aches (e.g., fibromyalgia), myopathy or myositis, whether or not it is related to treatment with statins or other lipid modifying drugs.
  * Renal impairment as defined by a calculated glomerular filtration rate < 60 mL/min
  * History of diabetes mellitus, or history of post-prandial and/or random blood glucose > 200 mg/dl or fasting glucose > 125 mg/dL or currently taking diabetes medications to manage fasting glucose levels (e.g., thiazolidinediones, sulfonylureas, insulin, metformin).
  * History of pancreatitis within 10 years of screening.
  * Any concurrent serious illness (e.g., severe chronic obstructive pulmonary disease, sleep apnea, history of malignancy other than skin cancer within 5 years of initial diagnosis or with evidence of recurrence) that may interfere with a subject from completing the study.
  * Current or chronic history of liver disease, or known hepatic or biliary abnormalities.
  * Active peptic ulcer disease and/or history of peptic ulcer disease or gastrointestinal bleeding within 12 months prior to screening.
  * History of kidney stones within 10 years of screening.
  * History of uncorrected thyroid dysfunction or an abnormal thyroid function test assessed by thyroid stimulating hormone (TSH) at Screening. (NOTE: subjects with hypothyroidism on a stable dose of thyroid replacement therapy for at least 3 months prior to screening and who have a screening TSH within the normal range may participate.)
  * Symptomatic cholelithiasis or obstructive or inflammatory gallbladder disease within 3 months prior to screening.
  * Gastrointestinal disease that could affect fat or bile acid absorption, or the pharmacokinetics or pharmacodynamics of the study drugs, including inflammatory bowel disease, chronic diarrhea, Crohn's disease or malabsorption syndromes within the past year.
  * Gastrointestinal surgery that may affect the pharmacokinetics or pharmacodynamics of the study drugs.

Note: Subjects may be enrolled in the study if they have had a cholecystectomy three or more months before the time of screening and are stable and asymptomatic.

* Subjects taking ezetimibe monotherapy, fibrates, bile acid binding resins, nicotinic acid or fat absorption inhibitors are not eligible for Parts A and B.
* For females a hemoglobin < 11.5g/dL, and for males a hemoglobin < 12.5g/dL.
* Current inadequately controlled hypertension (blood pressure >= 160mmHg systolic or >= 100mmHg diastolic at screening). If blood pressure medication is changed as a result of screening, blood pressure will be re-measured after 6 weeks and must again meet these criteria.
* Significant electrocardiogram (ECG) abnormalities, defined as follows:

Heart Rate < 50 and >100bpm PR Interval <120 and > 220ms QRS duration < 70 and >120ms QTC Interval (Bazett) > 450ms Or, has clinically significant rhythm abnormalities identified during 24-hour screening Holter assessment. Subjects with left bundle branch block are excluded from the study. Subjects with partial right bundle branch block may be considered for inclusion following consultation with the GlaxoSmithKline (GSK) Medical Monitor. Subjects with Wolf-Parkinson-White (WPW) syndrome are excluded from the study.

* Creatinine phosphokinase (CPK) >= 2x ULN at screening.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* The subject has a positive pre-study drug-of-abuse screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Subjects will be excluded if they require treatment with systemic corticosteroids.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to dosing.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of sensitivity or untoward reaction to the study medications (GSK1292263, atorvastatin or ezetimibe), or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* History of intolerance to statins.
* Any change in concomitant medication (including multivitamins, herbal remedies, dietary supplements, and over-the-counter medication) within six weeks prior to screening that is not approved by GSK.
* On a diet that may affect study outcomes, or any change in diet, exercise habits or smoking status within six weeks prior to screening or planned change during study (e.g., new exercise program) other than that in the dietary instructions in the Study Procedures Manual.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Where participation in study would result in donation of blood in excess of approximately 500mL within a 56 day period.
* Subject is mentally or legally incapacitated.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Pregnant females as determined by positive urine hCG test at screening or prior to dosing.
* Lactating females.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* Unwilling to abstain from caffeine-or xanthine-containing products from Day -2 until Day 15.
* Subject is either an immediate family member of a participating investigator, study coordinator, employee of an investigator; or is a member of the staff conducting the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2010-09-14 (Actual); Primary Completion 2011-06-29 (Actual); Study Completion 2011-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (18):
- United States (18):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Stockton, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Port Orange, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Berlin, New Jersey
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Renton, Washington

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=GPR113779

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 21 centers in the United States during the period 14 September 2010 to 29 June 2011. There were 6 total participants in Part A, then Part B started with total of 281 participants which flowed through the rest of the phases of the trial. Part B had washout phase and run-In phase followed by treatment phase.
Pre-assignment Details: Total 130 participants were randomized and received at least one dose of study drug in the treatment period phase. Part B Run-In excludes those participants randomized to monotherapy arms; that is, these participant counts are only those who were receiving Atorvastatin.
Groups:
- Part A: Four participants on 80 milligrams (mg) atorvastatin [either for >=4 weeks prior to screening (80 mg), or for 2 weeks, if the dose was escalated from a stable dose of 40mg], received GSK1292263 800 mg for 2 weeks, and 2 participants not on lipid-modifying treatment received GSK1282263 800 mg alone for 2 weeks.
- Part B Washout: Participants were washed off their prior lipid-lowering therapy for 4 weeks.
- Part B Run-in: Eligible participants were randomized to receive 10 mg open-labeled atorvastatin or 80 mg open-labeled atorvastatin for a 4-week stabilization run-in period.
- Part B Pooled Treatment Arm: In this pooled arm, after washout, randomized participants were stratified into 11 arms to receive either atorvastatin 10 mg along with 100 mg or 300 mg or 800 mg of GSK129226 or placebo or ezetimibe 10 mg once daily for 2 weeks; or atorvastatin 80 mg along with 800 mg of GSK129226 or placebo once daily for 2 weeks; or monotherapy (100 mg, 300 mg or 800 mg of GSK1292263 or placebo) once daily for 2 weeks.
Period: Part A
Arm/Group | Part A | Part B Washout | Part B Run-in | Part B Pooled Treatment Arm
Started | 6 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part B Washout
Arm/Group | Part A | Part B Washout | Part B Run-in | Part B Pooled Treatment Arm
Started | 0 | 281 | 0 | 0
Completed | 0 | 136 | 0 | 0
Not Completed | 0 | 145 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 14 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 14 | 0 | 0
Not completed — Reached defined stopping criteria | 0 | 2 | 0 | 0
Not completed — Did not meet continuation criteria | 0 | 112 | 0 | 0
Period: Part B Run-in
Arm/Group | Part A | Part B Washout | Part B Run-in | Part B Pooled Treatment Arm
Started | 0 | 0 | 89 | 0
Completed | 0 | 0 | 83 | 0
Not Completed | 0 | 0 | 6 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 0
Period: Part B Pooled Treatment Arm
Arm/Group | Part A | Part B Washout | Part B Run-in | Part B Pooled Treatment Arm
Started | 0 | 0 | 0 | 130
Completed | 0 | 0 | 0 | 127
Not Completed | 0 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: One participant was withdrawn prior to washout period. 34 participants did not complete washout phase. 111 participants did not qualify to continue in the study after completing the Washout Phase. 6 participants were withdrawn during run-in phase and 3 participants were withdrawn during treatment phase.
Groups:
- Part A: Four participants on 80 mg atorvastatin [either for >=4 weeks prior to screening (80 mg), or for 2 weeks, if the dose was escalated from a stable dose of 40 mg], received GSK1292263 800 mg for 2 weeks, and 2 participants not on lipid-modifying treatment received GSK1282263 800 mg alone for 2 weeks.
- Part B: Part B included Washout phase (Participants were washed off their prior lipid-lowering therapy for 4 weeks), Run-in phase (Eligible participants were randomized to receive 10 mg open-labeled atorvastatin or 80 mg open-labeled atorvastatin for a 4-week stabilization run-in period) and Treatment phase (Randomized participants after washout received monotherpy (100 mg, 300 mg or 800 mg of GSK1292263 or placebo) for 2 weeks. Participants in the 10mg atorvastatin run-in group received GSK1292263, 300 mg QD GSK1292263, 800 mg QD GSK1292263, placebo for GSK1292263 or 10 mg open-label ezetimibe for 2 weeks. Participants in the 80 mg atorvastatin run-in group received 800 mg QD GSK1292263 and placebo for GSK1292263 for 2 weeks)
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Total
Number analyzed (Participants) | 6 | 281 | 287
Age, Continuous [Mean (Standard Deviation); unit: Years] — Data is presented for Part A Population: N=6
  Years
    number analyzed (Participants) | 6 | 0 | 6
    (all) | 49.2 (5.34) |  | 49.2 (5.34)
Age, Continuous [Mean (Standard Deviation); unit: Years] — Data is presented for Part B Population: N=281
  Years
    number analyzed (Participants) | 0 | 281 | 281
    (all) |  | 57.7 (9.97) | 57.7 (9.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 152 | 152
  Male | 6 | 129 | 135
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 1 | 32 | 33
  American Indian or Alaska Native | 0 | 1 | 1
  Asian - Central/South Asian Heritage | 0 | 2 | 2
  Asian - Japanese Heritage | 0 | 2 | 2
  Asian - South East Asian Heritage | 0 | 1 | 1
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  White - Arabic/North African Heritage | 0 | 7 | 7
  White - White/Caucasian/European Heritage | 5 | 230 | 235
  White - Mixed Race | 0 | 1 | 1
  Mixed Race | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)- Part A
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, or is an important medical events that jeopardize the participants or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition, or a drug-induced liver injury.
Time Frame: Up to Day 26
Population: Safety Population consisted of all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- 80 mg Atorvastatin + 800 mg GSK1292263: Participants on 80 mg atorvastatin (either for >=4 weeks prior to screening (80 mg), or for 2 weeks, if the dose was escalated from a stable dose of 40 mg) received 800 mg of GSK1292263 for 2 weeks once daily immediately after eating the breakfast meal.
- 800 mg GSK1292263: Participants not on lipid-modifying treatment received GSK1282263 alone for 2 weeks once daily immediately after eating the breakfast meal.
Arm/Group | 80 mg Atorvastatin + 800 mg GSK1292263 | 800 mg GSK1292263
Number analyzed (Participants) | 4 | 2
Participants
  Any AE | 0 | 2
  Any SAE | 0 | 0

2. Primary Outcome: Number of Participants With Any AEs and SAEs- Part B (Washout)
Description: as for outcome 1
Time Frame: Up to Day 28
Population: All subject Population consisted of all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Pre-treatment: This was the time period prior to Day 1 of Washout Phase.
- Washout: During the 4 weeks washout period, participants were asked to stop their lipid-modifying drugs.
Arm/Group | Pre-treatment | Washout
Number analyzed (Participants) | 281 | 281
Participants
  Any AE | 14 | 37
  Any SAE | 0 | 0

3. Primary Outcome: Number of Participants With Any AEs and SAEs- Part B (Run-in)
Description: as for outcome 1
Time Frame: Up to Day 28
Population: All subject Population
Measure: Count of Participants; unit: Participants
Groups:
- Atorvastatin 10 mg: After washout participants received atorvastatin 10 mg for a 4-week stabilization Run-in Period.
- Atorvastatin 80 mg: After washout participants received atorvastatin 80 mg for a 4-week stabilization Run-in Period.
Arm/Group | Atorvastatin 10 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 62 | 27
Participants
  Any AE | 19 | 8
  Any SAE | 0 | 0

4. Primary Outcome: Number of Participants With Any AEs and SAEs- Part B (Pooled Treatment Arm)
Description: as for outcome 1
Time Frame: Up to Day 26
Population: All subject Population
Measure: Count of Participants; unit: Participants
Groups:
- Atorvastatin 10 mg + GSK1292263 100 mg: Participants received 10 mg atorvastatin along with GSK1292263 100 mg once daily for 2 weeks.
- Atorvastatin 10 mg + GSK1292263 300 mg: Participants received 10 mg atorvastatin along with GSK1292263 300 mg once daily for 2 weeks.
- Atorvastatin 10 mg + GSK1292263 800 mg: Participants received 10 mg atorvastatin along with GSK1292263 800 mg once daily for 2 weeks.
- Atorvastatin 10 mg + Placebo: Participants received 10 mg atorvastatin along with placebo matching to GSK1292263 once daily for 2 weeks.
- Atorvastatin 10 mg + Ezetimibe 10 mg: Participants received 10 mg atorvastatin along with Ezetimibe 10 mg once daily for 2 weeks.
- Atorvastatin 80 mg + GSK1292263 800 mg: Participants received 80 mg atorvastatin along with GSK1292263 800 mg once daily for 2 weeks.
- Atorvastatin 80 mg + Placebo: Participants received 80 mg atorvastatin along with placebo matching to GSK1292263 once daily for 2 weeks.
- GSK1292263 100 mg: After washout, participants were randomized to receive monotherapy of GSK1292263 100 mg once daily for 2 weeks
- GSK1292263 300 mg: After washout, participants were randomized to receive monotherapy of GSK1292263 300 mg once daily for 2 weeks
- GSK1292263 800 mg: After washout, participants were randomized to receive monotherapy of GSK1292263 800 mg once daily for 2 weeks
- Placebo: After washout, participants were randomized to receive placebo matching to GSK1292263 once daily for 2 weeks
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo | GSK1292263 100 mg | GSK1292263 300 mg | GSK1292263 800 mg | Placebo
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 13 | 12 | 13 | 11 | 12 | 13 | 11
Participants
  Any AE | 6 | 2 | 3 | 3 | 4 | 6 | 4 | 5 | 7 | 8 | 4
  Any SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal- Clinically Significant Electrocardiogram (ECG) Findings- Part A
Description: Single ECGs were taken after admission on Day -1 and at Follow-up (up to Day 26). On Days 1, 7, and 14 single ECGS were taken pre-breakfast (fasting) and at 1, 3, 6, 8, 14 and 24 hours post-dose. ECGs were taken in supine position. Additional ECGs were taken at the discretion of the investigator as needed based on symptoms or ECG findings. No value found to be abnormal clinically significant in Part A of the study.
Time Frame: Up to Day 26
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- Atorvastatin 80 mg + GSK1292263 800 mg: Participants on 80 mg atorvastatin (either for >=4 weeks prior to screening (80 mg), or for 2 weeks, if the dose was escalated from a stable dose of 40 mg) received 800 mg of GSK1292263 for 2 weeks once daily immediately after eating the breakfast meal.
- GSK1292263 800 mg: Participants not on lipid-modifying treatment received GSK1282263 alone for 2 weeks once daily immediately after eating the breakfast meal.
Arm/Group | Atorvastatin 80 mg + GSK1292263 800 mg | GSK1292263 800 mg
Number analyzed (Participants) | 4 | 2
Participants | 0 | 0

6. Primary Outcome: Number of Participants With Abnormal Clinically Significant ECG Findings- Part B (Washout)
Description: ECGs were taken at Screening, and on Day1 and Day 28. Single assessments were made. ECGs were taken in supine position. Additional ECGs were taken at the discretion of the investigator as needed based on symptoms or ECG findings.
Time Frame: Up to Day 28
Population: All subject Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Washout
Number analyzed (Participants) | 281
Participants
  Day 1 | 1
  Day 28: number analyzed (Participants) | 241
  Day 28 | 1

7. Primary Outcome: Number of Participants With Abnormal Clinically Significant ECG Findings- Part B (Run-in)
Description: ECGs were taken on Day 28. Single assessments were made. ECGs were taken in supine position. Additional ECGs were taken at the discretion of the investigator as needed based on symptoms or ECG findings. No data found to be abnormal clinically significant in run-in phase.
Time Frame: Day 28
Population: All subjects Population. Only those participants present during Run in/Day 28 were evaluated/included.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin 10 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 59 | 25
Participants | 0 | 0

8. Primary Outcome: Number of Participants With Abnormal Clinically Significant ECG Findings- Part B (Pooled Treatment Arm)
Description: Single ECGs were taken after admission on Day -2, and pre-breakfast on Days -1, 4, 10, and at Follow-up. On Days 1, 7, and 14 single ECGS were taken pre-breakfast (fasting) and at 1, 3, 6, 8, 14 and 24 hours post-dose. ECGs were taken in supine position. Additional ECGs were taken at the discretion of the investigator as needed based on symptoms or ECG findings. The data was found to be abnormal clinically significant in treatment phase.
Time Frame: Up to Day 26
Population: All subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo | GSK1292263 100 mg | GSK1292263 300 mg | GSK1292263 800 mg | Placebo
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 13 | 12 | 13 | 11 | 12 | 13 | 11
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance (PCI)- Part A
Description: Assessment of vital signs including systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate was performed after admission on Day -1 and at Follow-up. On Days 1, 7 and 14, they were taken at pre-dose, 1, 3, 6, 8, 14 and 24 hours after the morning dose. At each time point, assessment was performed after resting in a supine or semi-supine position for at least 10 minutes. Data for only those parameters are presented for which findings are of PCI either high or low.
Time Frame: Up to Day 26
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin 80 mg + GSK1292263 800 mg | GSK1292263 800 mg
Number analyzed (Participants) | 4 | 2
Participants
  DBP, high | 0 | 1
  DBP, low | 0 | 0

10. Primary Outcome: Number of Participants With Vital Signs of PCI- Part B (Washout)
Description: Assessment of vital signs including SBP, DBP heart rate was performed at Screening, on Days 1, 14 and 28 in the morning. At each time point, assessment was performed after resting in a supine or semi-supine position for at least 10 minutes. Data for only those parameters are presented for which findings are of PCI either high or low.
Time Frame: Up to day 28
Population: All subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Washout
Number analyzed (Participants) | 281
Participants
  SBP, high | 4
  Heart rate, high | 1

11. Primary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance- Part B (Run-in)
Description: Assessment of vital signs including SBP, DBP and heart rate was performed on Days 1, 14 and 28 in the morning. At each time point, assessment was performed after resting in a supine or semi-supine position for at least 10 minutes. Data for only those parameters are presented for which findings are of PCI either high or low.
Time Frame: Up to day 28
Population: All subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin 10 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 62 | 27
Participants
  SBP, high | 1 | 0
  SBP, low | 0 | 0

12. Primary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance- Part B (Pooled Treatment Arm)
Description: Assessment of vital signs including SBP, DBP and heart rate was performed after admission on Day-2, and pre-breakfast on Days -1, 4, and 10 in a fasting state early in the morning (prior to dosing), and at Follow-up. On Days 1, 7 and 14, they were also be taken at 1, 3, 6, 9, 12 and 24 hours after the morning dose. At each time point, assessment was performed after resting in a supine or semi-supine position for at least 10 minutes. Data for only those parameters are presented for which findings are of PCI either high or low.
Time Frame: Up to Day 26
Population: All subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo | GSK1292263 100 mg | GSK1292263 300 mg | GSK1292263 800 mg | Placebo
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 13 | 12 | 13 | 11 | 12 | 13 | 11
Participants
  SBP, high | 0 | 0 | 1 | 3 | 2 | 1 | 2 | 1 | 2 | 0 | 0
  DBP, high | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  DBP, low | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
  Heart rate, high | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Abnormal Hematology Value of PCI- Part A
Description: Blood samples were collected fasting on Day -1, and prior to breakfast (early in the morning, fasting) on Days 2, 4, 7, 11 and on Day 15 prior to checkout (24 hours post last-dose), and at Follow-up. When this resulted in multiple samples at the same time point, only one sample was collected (example, when 24 hours post-dose = pre-dose (time 0) for the next dose). Data for only those parameters (Hematocrit, Hemoglobin and Total neutrophils) are presented for which findings are of PCI either high or low.
Time Frame: Up to Day 26
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin 80 mg + GSK1292263 800 mg | GSK1292263 800 mg
Number analyzed (Participants) | 4 | 2
Participants
  Hematocrit, high | 2 | 1
  Hemoglobin, high | 2 | 0
  Total neutrophil, low | 1 | 0

14. Primary Outcome: Number of Participants With Abnormal Hematology Value of PCI- Part B (Washout)
Description: Blood samples were collected at screening, and on Days 1 (first day of washout), 14 and 28 prior to breakfast (early in the morning, fasting). Data for only those parameters (White blood cells [WBC], Total neutrophils, Hematocrit and Lymphocytes) are presented for which findings are of PCI either high or low.
Time Frame: Up to Day 28
Population: All subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Washout
Number analyzed (Participants) | 281
Participants
  WBC, high | 1
  WBC, low | 1
  Total neutrophil, low | 1
  Hematocrit, high | 2
  Lymphocytes, low | 2

15. Primary Outcome: Number of Participants With Abnormal Hematology Value of PCI- Part B (Run-in)
Description: Blood samples were collected on Day 14 and 28 prior to breakfast (early in the morning, fasting). Data for only those parameters (Lymphocytes) are presented for which findings are of PCI either high or low.
Time Frame: Days 14 and 28
Population: All subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin 10 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 62 | 27
Participants
  Lymphocytes, low | 0 | 1
  Lymphocytes, high | 0 | 0

16. Primary Outcome: Number of Participants With Abnormal Hematology Value of PCI- Part B (Pooled Treatment Arm)
Description: Blood samples were collected fasting on Day -2, and prior to breakfast (early in the morning, fasting) on Days 2 (pre-dose), 4, 7, 10, 13 and on Day 15 prior to checkout (24hrs post-dose), and at Follow-up. When this resulted in multiple samples at the same time point, only one sample was collected (example, when 24hrs post dose = pre-dose (time 0) for the next dose). Data for only those parameters (Platelet count, Total neutrophils and Lymphocytes) are presented for which findings are of PCI either high or low.
Time Frame: Up to Day 26
Population: All subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo | GSK1292263 100 mg | GSK1292263 300 mg | GSK1292263 800 mg | Placebo
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 13 | 12 | 13 | 11 | 12 | 13 | 11
Participants
  Platelet count, low | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Total neutrophils, low | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocytes, low | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0

17. Primary Outcome: Number of Participants With Abnormal Clinical Chemistry Value of PCI- Part A
Description: Samples were collected fasting on Day -1, and prior to breakfast (early in the morning, fasting) on Days 2, 4, 7, 11 and on Day 15 prior to checkout (24 hours post last-dose), and at Follow-up. When this resulted in multiple samples at the same time point, only one sample was collected (example, when 24 hours post-dose = pre-dose (time 0) for the next dose). No parameter was found to have any value of PCI.
Time Frame: Up to Day 26
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin 80 mg + GSK1292263 800 mg | GSK1292263 800 mg
Number analyzed (Participants) | 4 | 2
Participants | 0 | 0

18. Primary Outcome: Number of Participants With Abnormal Clinical Chemistry Value of PCI- Part B (Washout)
Description: Samples were collected at screening, and on Days1 (first day of washout), 14 and 28 prior to breakfast (early in the morning, fasting). Data for only those parameters (Inorganic phosphorus, Sodium, Alanine aminotransferase [ALT], Potassium, Creatinine, Calcium, magnesium, Glucose, Total Bilirubin, Carbon dioxide/bicarbonate [CO2/HCO3] and Aspartate aminotransferase [AST]) are presented for which findings are of PCI either high or low.
Time Frame: Up to Day 28
Population: All subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Washout
Number analyzed (Participants) | 281
Participants
  Inorganic phosphorus, high | 3
  Inorganic phosphorus, low | 2
  Sodium, high | 1
  Sodium, low | 1
  ALT, high | 3
  Potassium, high | 3
  Potassium, low | 1
  Creatinine, high | 1
  Calcium, high | 2
  Magnesium, high | 32
  Glucose, high | 4
  Glucose, low | 1
  Total bilirubin, high | 6
  CO2/bicarbonate, low | 1
  AST, high | 1

19. Primary Outcome: Number of Participants With Abnormal Clinical Chemistry Value of PCI- Part B (run-in)
Description: Samples were collected on Day 14 and 28 prior to breakfast (early in the morning, fasting). Data for only those parameters (Glucose, Magnesium, ALT, AST, Calcium, Inorganic phosphorus and Total bilirubin) are presented for which findings are of PCI either high or low.
Time Frame: Days 14 and 28
Population: All subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin 10 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 62 | 27
Participants
  Glucose, high | 1 | 0
  Magnesium, high | 5 | 5
  ALT, high | 1 | 0
  AST, high | 1 | 0
  Calcium, high | 0 | 1
  Inorganic phosphorus, low | 0 | 1
  Total bilirubin, high | 0 | 1

20. Primary Outcome: Number of Participants With Abnormal Clinical Chemistry Value of PCI- Part B (Pooled Treatment Arm)
Description: Samples were collected fasting on Day -2, and prior to breakfast (early in the morning, fasting) on Days 2 (pre-dose), 4, 7, 10, 13 and on Day 15 prior to checkout (24 hours post-dose), and at Follow-up. When this resulted in multiple samples at the same time point, only one sample was collected (example, when 24 hours post dose = pre-dose (time 0) for the next dose). Data for only those parameters (Glucose, Total bilirubin, Albumin, Magnesium, CO2/HCO3, Calcium, ALT, AST, Inorganic phosphorus, Potassium and Sodium) are presented for which findings are of PCI either high or low.
Time Frame: Up to Day 26
Population: All subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo | GSK1292263 100 mg | GSK1292263 300 mg | GSK1292263 800 mg | Placebo
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 13 | 12 | 13 | 11 | 12 | 13 | 11
Participants
  Glucose, high | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Glucose, low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Total bilirubin, high | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
  Albumin, low | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Magnesium, high | 0 | 1 | 2 | 1 | 1 | 2 | 3 | 2 | 3 | 2 | 2
  CO2/HCO3, high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  CO2/HCO3, low | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, high | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Calcium, low | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  ALT, high | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST, high | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Inorganic phosphorus, high | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Sodium, high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

21. Primary Outcome: Maximum Observed Concentration (Cmax) of GSK1292263- Part A
Description: Serial blood samples for the determination of the PK for GSK1292263 on Days 1 and 14 were collected at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hours post-morning dose (no 48 hour sample on Day 1).
Time Frame: On Days 1 and 14 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hours post-morning dose
Population: Pharmacokinetic (PK) Parameter Population was defined as participants in the 'PK Concentration' population for whom PK parameters were derived. The 'PK Concentration Population' was defined as participants in the 'All Subjects' Population for whom a PK sample was obtained and analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Atorvastatin 80 mg + GSK1292263 800 mg | GSK1292263 800 mg
Number analyzed (Participants) | 4 | 2
nanograms per milliliter
  Day 1 | 976.335 (16.6353) | 986.811 (46.4825)
  Day 14 | 1118.344 (20.6141) | 948.764 (6.5356)

22. Primary Outcome: Cmax of GSK1292263- Part B (Pooled Treatment Arm)
Description: For co-dosing arms, serial blood samples for the determination of the PK of GSK1292263 were taken on Days 1 and 14. For monotherapy arms, serial blood samples for the determination of the PK of GSK1292263 were collected on Days 1 and 14. Blood samples for PK were collected on Day 1 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, and 24 hours post-morning dose. Blood samples for PK were collected on Day 14 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hours post-morning dose (48 hours PK sample was collected on Day 16).
Time Frame: On Day 1 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, and 24 hours post-morning dose. On Day 14 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hours post-morning dose
Population: PK parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 80 mg + GSK1292263 800 mg | GSK1292263 100 mg | GSK1292263 300 mg | GSK1292263 800 mg
Number analyzed (Participants) | 7 | 7 | 11 | 12 | 11 | 12 | 13
nanograms per milliliter
  Day 1: number analyzed (Participants) | 5 | 6 | 8 | 12 | 11 | 12 | 12
  Day 1 | 281.321 (35.9671) | 475.297 (36.5131) | 808.278 (20.0646) | 790.315 (32.5080) | 263.279 (43.0140) | 478.676 (21.2079) | 787.922 (36.7864)
  Day 14: number analyzed (Participants) | 6 | 7 | 7 | 11 | 10 | 12 | 13
  Day 14 | 361.595 (25.9981) | 639.687 (33.6608) | 886.418 (31.3931) | 848.082 (25.1892) | 364.936 (39.1918) | 590.949 (20.7601) | 782.914 (81.2992)

23. Primary Outcome: Time of Occurrence of Cmax (Tmax) and Terminal Phase Half-life (t1/2) GSK1292263- Part A
Description: Serial blood samples for the determination of the PK for GSK1292263, on Days 1 and 14 were collected at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hours post-morning dose (no 48 hour sample on Day 1).
Time Frame: as for outcome 21
Population: PK parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Atorvastatin 80 mg + GSK1292263 800 mg | GSK1292263 800 mg
Number analyzed (Participants) | 4 | 2
hours
  tmax, Day 1 | 6.000 [4.00 to 8.00] | 5.000 [4.00 to 6.00]
  tmax, Day 14 | 3.000 [3.00 to 4.00] | 5.067 [4.00 to 6.13]
  t1/2, Day 1: number analyzed (Participants) | 3 | 1
  t1/2, Day 1 | 11.185 [8.81 to 11.61] | 16.164 [16.164 to 16.164]
  t1/2, Day 14 | 20.629 [13.76 to 28.80] | 19.395 [16.54 to 22.25]

24. Primary Outcome: Lag Time Before Observation of Drug Concentrations in Sampled Matrix (Tlag) of GSK1292263- Part A
Description: Serial blood samples for the determination of the PK for GSK1292263 on Days 1 were collected at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hours post-morning dose (no 48h sample on Day 1).
Time Frame: On Day 1 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hours post-morning dose
Population: PK parameter Population
Measure: Median (Full Range); unit: hours
Arm/Group | Atorvastatin 80 mg + GSK1292263 800 mg | GSK1292263 800 mg
Number analyzed (Participants) | 4 | 2
hours | 0.250 [0.00 to 0.50] | 0.000 [0.00 to 0.00]

25. Primary Outcome: Tmax and t1/2 of GSK1292263- Part B (Pooled Treatment Arm)
Description: as for outcome 22
Time Frame: as for outcome 22
Population: PK parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 80 mg + GSK1292263 800 mg | GSK1292263 100 mg | GSK1292263 300 mg | GSK1292263 800 mg
Number analyzed (Participants) | 7 | 7 | 11 | 12 | 11 | 12 | 13
hours
  tmax, Day 1: number analyzed (Participants) | 5 | 6 | 8 | 12 | 11 | 12 | 12
  tmax, Day 1 | 3.983 [3.00 to 6.00] | 5.008 [3.98 to 8.00] | 4.000 [4.00 to 8.33] | 4.000 [3.98 to 8.08] | 4.000 [1.50 to 8.00] | 4.000 [2.00 to 8.00] | 3.475 [1.98 to 7.97]
  tmax, Day 14: number analyzed (Participants) | 6 | 7 | 6 | 11 | 10 | 12 | 13
  tmax, Day 14 | 5.000 [0.83 to 8.00] | 4.000 [2.08 to 4.02] | 4.000 [1.50 to 4.05] | 4.000 [1.50 to 4.00] | 4.000 [3.98 to 6.00] | 3.983 [1.98 to 6.00] | 4.000 [0.43 to 5.98]
  t1/2, Day 1: number analyzed (Participants) | 1 | 3 | 4 | 4 | 7 | 5 | 1
  t1/2, Day 1 | 12.630 [12.63 to 12.63] | 10.270 [6.07 to 10.55] | 10.416 [9.29 to 26.11] | 12.372 [6.72 to 23.08] | 15.305 [12.25 to 21.78] | 14.342 [13.38 to 20.30] | 14.464 [14.464 to 14.464]
  t1/2, Day 14: number analyzed (Participants) | 6 | 6 | 5 | 7 | 9 | 10 | 11
  t1/2, Day 14 | 26.453 [17.02 to 163.25] | 21.569 [15.73 to 37.15] | 21.846 [10.52 to 36.52] | 24.225 [16.86 to 34.21] | 23.893 [17.43 to 43.62] | 25.203 [10.67 to 62.63] | 19.478 [12.40 to 67.78]

26. Primary Outcome: Tlag of GSK1292263- Part B (Pooled Treatment Arm)
Description: Blood samples for PK were collected on Day 1 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, and 24 hours post-morning dose.
Time Frame: On Day 1 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, and 24 hours post-morning dose.
Population: PK parameter Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 80 mg + GSK1292263 800 mg | GSK1292263 100 mg | GSK1292263 300 mg | GSK1292263 800 mg
Number analyzed (Participants) | 5 | 6 | 8 | 12 | 11 | 12 | 12
hours | 0.000 [0.00 to 0.50] | 0.000 [0.00 to 0.50] | 0.000 [0.00 to 1.03] | 0.000 [0.00 to 0.50] | 0.000 [0.00 to 1.03] | 0.000 [0.00 to 1.00] | 0.000 [0.00 to 0.50]

27. Primary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to 24 Hours [AUC(0-24)] of GSK1292263- Part A
Description: as for outcome 23
Time Frame: as for outcome 21
Population: PK parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms hour per milliliter
Arm/Group | Atorvastatin 80 mg + GSK1292263 800 mg | GSK1292263 800 mg
Number analyzed (Participants) | 4 | 2
nanograms hour per milliliter
  Day 1: number analyzed (Participants) | 3 | 1
  Day 1 | 12953.89 (16.976) | 12032.21 (NA) — Only one participant was analyzed.
  Day 14 | 13206.52 (15.070) | 11890.40 (5.730)

28. Primary Outcome: AUC(0-24) of GSK1292263- Part B (Pooled Treatment Arm)
Description: as for outcome 22
Time Frame: as for outcome 22
Population: PK parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms hour per milliliter
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 80 mg + GSK1292263 800 mg | GSK1292263 100 mg | GSK1292263 300 mg | GSK1292263 800 mg
Number analyzed (Participants) | 7 | 7 | 11 | 12 | 11 | 12 | 13
nanograms hour per milliliter
  Day 1: number analyzed (Participants) | 4 | 5 | 7 | 9 | 8 | 8 | 8
  Day 1 | 4218.02 (54.264) | 5373.78 (64.021) | 10384.24 (15.165) | 9812.21 (25.708) | 2753.61 (48.535) | 5342.77 (18.108) | 8937.99 (21.080)
  Day 14: number analyzed (Participants) | 6 | 7 | 7 | 11 | 10 | 11 | 13
  Day 14 | 4968.29 (24.683) | 7484.67 (51.772) | 11224.58 (44.087) | 10760.74 (22.081) | 4061.78 (35.242) | 6737.82 (28.082) | 8837.31 (79.003)

29. Primary Outcome: Trough Concentration of GSK1292263
Description: Trough samples for GSK1292263 PK (all treatment arms) were planned to be collected early in the morning on Days 13, 14, 15 and 16 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hours post-morning dose (48h PK sample was collected on Day 16). (pre-dose for Days 13 and 14; trough Day 15 = 24h post last dose; trough Day 16 = 48h post last dose).
Time Frame: On Days 13, 14, 15 and 16 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hours post-morning dose
Population: PK concentration Population. Data was not collected for this outcome measure.
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 80 mg + GSK1292263 800 mg | GSK1292263 100 mg | GSK1292263 300 mg | GSK1292263 800 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

30. Primary Outcome: Cmax of Atorvastatin- Part A
Description: Serial blood samples for the determination of the PK for atorvastatin on Day -1 was collected at immediately pre-morning dose=pre-breakfast (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14 and 24 hours post-morning dose (24 hour sample Day -1 = 0 hour sample Day 1). Serial blood samples for the determination of the PK for atorvastatin on Days 1 and 14 will be collected at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hour post-morning dose (no 48h sample on Day 1).
Time Frame: On Day -1 at immediately pre-morning dose=pre-breakfast (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14 and 24 hours post-morning dose. on Days 1 and 14 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hour post-morning dose.
Population: PK parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Atorvastatin 80 mg + GSK1292263 800 mg
Number analyzed (Participants) | 4
nanograms per milliliter
  Day -1 | 45.587 (130.4168)
  Day 1 | 25.867 (88.8156)
  Day 14 | 38.443 (71.1418)

31. Primary Outcome: Cmax of Atorvastatin- Part B (Pooled Treatment Arm)
Description: For co-dosing arms, serial blood samples for the determination of the PK of atorvastatin were collected on Day -1 and for atorvastatin on Days 1 and 14. Blood samples for PK were collected on Days -1 (co-dosing arms only) and 1 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, and 24 hours post-morning dose. Blood samples for PK were collected on Day 14 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hours post-morning dose (48 hour PK sample was collected on Day 16).
Time Frame: On Days -1 and 1 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, and 24 hours post-morning dose. on Day 14 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hours post-morning dose
Population: PK parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo
Number analyzed (Participants) | 7 | 7 | 11 | 12 | 6 | 12 | 13
nanograms per milliliter
  Day -1: number analyzed (Participants) | 4 | 5 | 10 | 12 | 6 | 12 | 13
  Day -1 | 2.045 (41.3980) | 2.454 (34.6820) | 1.683 (54.1388) | 1.816 (54.6608) | 2.003 (73.2912) | 42.376 (113.1276) | 37.058 (47.5590)
  Day 1: number analyzed (Participants) | 4 | 5 | 11 | 12 | 5 | 12 | 13
  Day 1 | 1.292 (26.6345) | 2.195 (47.6989) | 1.926 (47.0899) | 1.852 (57.6472) | 1.872 (64.1762) | 31.018 (81.5136) | 45.781 (38.4790)
  Day 14: number analyzed (Participants) | 4 | 5 | 10 | 12 | 5 | 11 | 13
  Day 14 | 1.453 (14.5258) | 2.154 (69.0856) | 2.139 (74.2524) | 1.640 (68.6754) | 1.949 (56.7747) | 38.419 (71.2059) | 41.092 (73.0152)

32. Primary Outcome: Tmax of Atorvastatin- Part A
Description: as for outcome 30
Time Frame: as for outcome 30
Population: PK parameter Population.
Measure: Median (Full Range); unit: hours
Arm/Group | Atorvastatin 80 mg + GSK1292263 800 mg
Number analyzed (Participants) | 4
hours
  Day -1 | 3.000 [0.50 to 4.00]
  Day 1 | 4.000 [3.00 to 6.00]
  Day 14 | 2.250 [1.00 to 3.00]

33. Primary Outcome: Tmax of Atorvastatin- Part B (Pooled Treatment Arm)
Description: as for outcome 31
Time Frame: as for outcome 31
Population: PK parameter Population. Only those participants available at specified time points were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo
Number analyzed (Participants) | 7 | 7 | 11 | 12 | 6 | 12 | 13
hours
  Day -1: number analyzed (Participants) | 4 | 5 | 10 | 12 | 6 | 12 | 13
  Day -1 | 2.500 [0.50 to 6.08] | 3.000 [1.50 to 6.00] | 3.983 [0.50 to 5.97] | 3.017 [0.50 to 6.08] | 4.000 [3.00 to 4.00] | 2.508 [0.50 to 6.00] | 1.517 [0.50 to 4.00]
  Day 1: number analyzed (Participants) | 4 | 5 | 11 | 12 | 5 | 12 | 13
  Day 1 | 4.992 [3.98 to 6.00] | 6.000 [3.95 to 6.00] | 3.000 [0.50 to 8.33] | 3.992 [1.50 to 6.08] | 4.000 [2.00 to 4.00] | 3.492 [1.03 to 6.03] | 2.000 [0.50 to 4.00]
  Day 14: number analyzed (Participants) | 4 | 5 | 10 | 12 | 5 | 11 | 13
  Day 14 | 4.000 [2.83 to 6.00] | 4.000 [3.00 to 6.00] | 3.500 [1.50 to 6.08] | 3.525 [1.50 to 6.00] | 2.000 [1.00 to 3.00] | 2.067 [0.50 to 5.93] | 3.000 [1.00 to 6.05]

34. Primary Outcome: AUC (0-24) of Atorvastatin- Part A
Description: as for outcome 31
Time Frame: as for outcome 31
Population: PK parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms hour per milliliter
Arm/Group | Atorvastatin 80 mg + GSK1292263 800 mg
Number analyzed (Participants) | 4
nanograms hour per milliliter
  Day -1 | 219.27 (77.893)
  Day 1 | 199.15 (73.974)
  Day 14 | 187.25 (52.566)

35. Primary Outcome: AUC (0-24) of Atorvastatin- Part B (Pooled Treatment Arm)
Description: as for outcome 31
Time Frame: as for outcome 31
Population: PK parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms hour per milliliter
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo
Number analyzed (Participants) | 7 | 7 | 11 | 12 | 6 | 12 | 13
nanograms hour per milliliter
  Day -1: number analyzed (Participants) | 4 | 5 | 10 | 12 | 5 | 11 | 12
  Day -1 | 23.16 (18.115) | 28.78 (26.611) | 19.26 (54.767) | 18.77 (51.122) | 19.59 (47.952) | 188.88 (70.744) | 173.62 (31.333)
  Day 1: number analyzed (Participants) | 4 | 5 | 11 | 12 | 5 | 11 | 13
  Day 1 | 17.84 (35.028) | 26.19 (30.561) | 20.83 (50.427) | 19.33 (55.620) | 19.05 (48.448) | 174.13 (55.829) | 186.73 (35.837)
  Day 14: number analyzed (Participants) | 4 | 5 | 9 | 12 | 4 | 11 | 12
  Day 14 | 15.58 (14.934) | 23.77 (38.501) | 20.41 (70.602) | 18.60 (56.102) | 20.24 (41.371) | 174.93 (59.199) | 188.31 (54.020)

36. Primary Outcome: Trough Concentration of Atorvastatin
Description: For co-dosing arms, serial blood samples for the determination of the PK of atorvastatin were planned to be collected on Day -1 and for atorvastatin on Days 1 and 14. Blood samples for PK were planned to be collected on Days -1 (co-dosing arms only) and 1 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, and 24 hours post-morning dose. Blood samples for PK were planned to be collected on Day 14 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hours post-morning dose (48 hour PK sample was planned to be collected on Day 16).
Time Frame: as for outcome 31
Population: PK parameter Population. Data was not collected for this outcome measure.
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

37. Primary Outcome: Percent Change From Baseline for Lipid Metabolism: Apolipoprotein A1 and Apolipoprotein B100 at Day 14
Description: Blood samples were collected fasting on Days 1 (pre-dose), 7 and 15 prior to checkout (24 hours post-dose), and at Follow-up. When this results in multiple samples at the same time point, only one sample will be collected (example, when 24 hours post-dose = pre-dose (time 0) for the next dose). Baseline was the closest scheduled value prior to dosing. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. If either the Baseline or post-randomization value is missing, the change from Baseline was set to missing as well. Percent change from Baseline was calculated as the change from Baseline divided by the Baseline value then multiplied by 100.
Time Frame: Baseline and Day 14
Population: All subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo | GSK1292263 100 mg | GSK1292263 300 mg | GSK1292263 800 mg | Placebo
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 13 | 12 | 13 | 11 | 12 | 13 | 11
Percent change
  Apolipoprotein A1, 24 hours: number analyzed (Participants) | 10 | 10 | 10 | 12 | 11 | 11 | 13 | 10 | 12 | 13 | 10
  Apolipoprotein A1, 24 hours | -1.93 (27.152) | -8.72 (31.791) | 4.17 (38.410) | -7.19 (27.383) | -3.88 (26.818) | -1.00 (35.805) | -5.81 (47.800) | 3.76 (41.281) | 29.90 (99.331) | -0.15 (39.226) | -0.18 (49.478)
  Apolipoprotein B100, 24 hours: number analyzed (Participants) | 10 | 10 | 10 | 12 | 13 | 11 | 13 | 10 | 12 | 13 | 11
  Apolipoprotein B100, 24 hours | 2.85 (31.217) | -17.93 (19.839) | -22.22 (20.393) | -5.03 (19.932) | -15.49 (13.681) | -27.08 (14.132) | 4.25 (27.890) | -10.21 (22.072) | -7.62 (23.573) | -10.95 (23.811) | -2.39 (15.932)
Statistical Analysis 1: Comparison: Atorvastatin 10 mg + GSK1292263 100 mg vs Placebo; Atorvastatin 10 mg + GSK1292263 100 mg vs Placebo: Apolipoprotein A1; Test type: Superiority or Other; Mean Difference (Net) = 5.473, 95% CI 2-sided [-15.7096 to 26.6553] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 2: Comparison: Atorvastatin 10 mg + GSK1292263 300 mg vs Placebo; Atorvastatin 10 mg + GSK1292263 300 mg vs Placebo: Apolipoprotein A1; Test type: Superiority or Other; Mean Difference (Net) = -0.598, 95% CI 2-sided [-21.7840 to 20.5888] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 3: Comparison: Atorvastatin 10 mg + GSK1292263 800 mg vs Placebo; Atorvastatin 10 mg + GSK1292263 800 mg vs Placebo: Apolipoprotein A1; Test type: Superiority or Other; Mean Difference (Net) = 11.906, 95% CI 2-sided [-9.3489 to 33.1602] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 4: Comparison: Atorvastatin 10 mg + Ezetimibe 10 mg vs Placebo; Atorvastatin 10 mg + Ezetimibe 10 mg vs Placebo: Apolipoprotein A1; Test type: Superiority or Other; Mean Difference (Net) = 3.671, 95% CI 2-sided [-16.9957 to 24.3384] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 5: Comparison: Atorvastatin 80 mg + GSK1292263 800 mg vs Placebo; Atorvastatin 80 mg + GSK1292263 800 mg vs Placebo: Apolipoprotein A1; Test type: Superiority or Other; Mean Difference (Net) = 4.618, 95% CI 2-sided [-28.2069 to 37.4425] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 6: Comparison: GSK1292263 100 mg vs Placebo; GSK1292263 100 mg vs Placebo: Apolipoprotein A1; Test type: Superiority or Other; Mean Difference (Net) = 7.713, 95% CI 2-sided [-17.0405 to 39.8527] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 7: Comparison: GSK1292263 300 mg vs Placebo; GSK1292263 300 mg vs Placebo: Apolipoprotein A1; Test type: Superiority or Other; Mean Difference (Net) = 1.934, 95% CI 2-sided [-21.0153 to 31.5504] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 8: Comparison: GSK1292263 800 mg vs Placebo; GSK1292263 800 mg vs Placebo: Apolipoprotein A1; Test type: Superiority or Other; Mean Difference (Net) = -2.466, 95% CI 2-sided [-23.7517 to 24.7608] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 9: Comparison: Atorvastatin 10 mg + GSK1292263 100 mg vs Placebo; Atorvastatin 10 mg + GSK1292263 100 mg vs Placebo: Apolipoprotein B100; Test type: Superiority or Other; Mean Difference (Net) = 13.743, 95% CI 2-sided [-3.2460 to 33.7161] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 10: Comparison: Atorvastatin 10 mg + GSK1292263 300 mg vs Placebo; Atorvastatin 10 mg + GSK1292263 300 mg vs Placebo: Apolipoprotein B100; Test type: Superiority or Other; Mean Difference (Net) = -7.428, 95% CI 2-sided [-21.3243 to 8.9224] — Statistical analysis was performed using LS mean value Atorvastatin
Statistical Analysis 11: Comparison: Atorvastatin 10 mg + GSK1292263 800 mg vs Placebo; Atorvastatin 10 mg + GSK1292263 800 mg vs Placebo: Apolipoprotein B100; Test type: Superiority or Other; Mean Difference (Net) = -13.960, 95% CI 2-sided [-26.8137 to 1.1513] — Statistical analysis was performed using LS mean value Atorvastatin
Statistical Analysis 12: Comparison: Atorvastatin 10 mg + Ezetimibe 10 mg vs Placebo; Atorvastatin 10 mg + Ezetimibe 10 mg vs Placebo: Apolipoprotein B100; Test type: Superiority or Other; Mean Difference (Net) = -2.903, 95% CI 2-sided [-16.6557 to 13.1191] — Statistical analysis was performed using LS mean value Atorvastatin
Statistical Analysis 13: Comparison: Atorvastatin 80 mg + GSK1292263 800 mg vs Placebo; Atorvastatin 80 mg + GSK1292263 800 mg vs Placebo: Apolipoprotein B100; Test type: Superiority or Other; Mean Difference (Net) = -28.231, 95% CI 2-sided [-45.1045 to -11.3579] — Statistical analysis was performed using LS mean value Atorvastatin
Statistical Analysis 14: Comparison: GSK1292263 100 mg vs Placebo; GSK1292263 100 mg vs Placebo: Apolipoprotein B100; Test type: Superiority or Other; Mean Difference (Net) = -6.100, 95% CI 2-sided [-23.5021 to 11.3014] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 15: Comparison: GSK1292263 300 mg vs Placebo; GSK1292263 300 mg vs Placebo: Apolipoprotein B100; Test type: Superiority or Other; Mean Difference (Net) = -8.490, 95% CI 2-sided [-25.2721 to 8.2918] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 16: Comparison: GSK1292263 800 mg vs Placebo; GSK1292263 800 mg vs Placebo: Apolipoprotein B100; Test type: Superiority or Other; Mean Difference (Net) = -9.687, 95% CI 2-sided [-26.0247 to 6.6498] — Statistical analysis was performed using LS mean value of GSK1292263

38. Primary Outcome: Percent Change From Baseline in Lipid Metabolism: Apolipoprotein E at Day 14 (24 Hours)
Description: as for outcome 37
Time Frame: Baseline and Day 14
Population: All subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Perecent change
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo | GSK1292263 100 mg | GSK1292263 300 mg | GSK1292263 800 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 12 | 13 | 11 | 13 | 10 | 12 | 13 | 11
Perecent change | -21.97 (16.373) | -3.92 (29.382) | -31.41 (17.369) | 34.28 (141.042) | -12.27 (42.191) | -13.19 (19.202) | -13.41 (30.613) | 1.35 (46.155) | -21.98 (37.910) | -33.75 (16.915) | -1.58 (36.044)
Statistical Analysis 1: Comparison: Atorvastatin 10 mg + GSK1292263 100 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -19.471, 95% CI 2-sided [-47.9323 to 3.2020] — Statistical analysis was performed using LS mean value Atorvastatin
Statistical Analysis 2: Comparison: Atorvastatin 10 mg + GSK1292263 300 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -5.910, 95% CI 2-sided [-38.1027 to 25.3126] — Statistical analysis was performed using LS mean value Atorvastatin
Statistical Analysis 3: Comparison: Atorvastatin 10 mg + GSK1292263 800 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -25.985, 95% CI 2-sided [-45.5492 to 1.8605] — Statistical analysis was performed using LS mean value Atorvastatin
Statistical Analysis 4: Comparison: Atorvastatin 10 mg + Ezetimibe 10 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -16.697, 95% CI 2-sided [-45.0846 to 13.3024] — Statistical analysis was performed using LS mean value Atorvastatin
Statistical Analysis 5: Comparison: Atorvastatin 80 mg + GSK1292263 800 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -6.036, 95% CI 2-sided [-27.2281 to 15.1569] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 6: Comparison: GSK1292263 100 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = 0.198, 95% CI 2-sided [-24.2901 to 32.6057] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 7: Comparison: GSK1292263 300 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -22.117, 95% CI 2-sided [-40.4767 to 1.9060] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 8: Comparison: GSK1292263 800 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -32.798, 95% CI 2-sided [-48.3842 to -12.5064] — Statistical analysis was performed using LS mean value of GSK1292263

39. Primary Outcome: Percent Change From Baseline in Lipid Metabolism: High Density Lipids Cholesterol (HDLc), Low Density Lipids Cholesterol (LDLc), Tryglycerides, Non-HDLc and Total Cholesterol at Day 14 (24 Hours)
Description: as for outcome 37
Time Frame: Baseline and Day 14
Population: All subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo | GSK1292263 100 mg | GSK1292263 300 mg | GSK1292263 800 mg | Placebo
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 13 | 12 | 13 | 11 | 12 | 13 | 11
Percent change
  HDLc: number analyzed (Participants) | 11 | 11 | 10 | 12 | 13 | 11 | 12 | 10 | 11 | 13 | 10
  HDLc | 7.50 (13.639) | 14.97 (7.700) | 31.09 (11.966) | -0.03 (14.714) | 6.03 (11.850) | 26.22 (15.840) | 4.50 (10.936) | 9.17 (10.277) | 9.76 (17.160) | 18.95 (12.847) | -1.37 (7.140)
  LDLc: number analyzed (Participants) | 11 | 11 | 10 | 12 | 13 | 11 | 12 | 10 | 11 | 13 | 10
  LDLc | -6.80 (14.522) | -10.01 (21.231) | -24.09 (18.017) | -0.37 (19.794) | -24.81 (12.317) | -18.63 (16.534) | 15.01 (59.194) | -10.24 (11.438) | -11.86 (16.873) | -19.94 (10.688) | 0.77 (11.347)
  Triglyceides: number analyzed (Participants) | 11 | 11 | 10 | 12 | 13 | 11 | 12 | 10 | 11 | 13 | 10
  Triglyceides | -18.67 (16.693) | -15.98 (24.307) | -32.81 (21.249) | 10.70 (32.177) | -10.44 (21.628) | -21.39 (28.190) | 2.27 (17.025) | -3.95 (23.855) | -30.84 (11.753) | -34.66 (21.197) | 18.90 (18.225)
  Non-HDLc: number analyzed (Participants) | 11 | 11 | 10 | 12 | 13 | 11 | 12 | 10 | 11 | 13 | 10
  Non-HDLc | -9.53 (8.502) | -11.67 (18.562) | -26.59 (13.742) | 2.08 (16.176) | -21.19 (11.920) | -21.88 (11.157) | -0.94 (8.977) | -9.32 (13.107) | -17.02 (12.376) | -22.62 (10.290) | 3.17 (9.283)
  Total cholesterol: number analyzed (Participants) | 11 | 11 | 10 | 12 | 13 | 11 | 12 | 10 | 11 | 13 | 10
  Total cholesterol | -5.17 (9.210) | -3.61 (12.355) | -10.31 (8.912) | 0.89 (12.671) | -14.23 (9.640) | -5.52 (7.721) | 1.09 (6.724) | -5.81 (10.091) | -12.06 (9.650) | -14.05 (7.614) | 2.18 (7.900)
Statistical Analysis 1: Comparison: Atorvastatin 10 mg + GSK1292263 100 mg vs Placebo; For HDLc; Test type: Superiority or Other; Mean Difference (Net) = 5.101, 95% CI 2-sided [-4.5469 to 14.7495] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 2: Comparison: Atorvastatin 10 mg + GSK1292263 300 mg vs Placebo; Fo HDLc; Test type: Superiority or Other; Mean Difference (Net) = 12.273, 95% CI 2-sided [2.5937 to 21.9532] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 3: Comparison: Atorvastatin 10 mg + GSK1292263 800 mg vs Placebo; For HDLc; Test type: Superiority or Other; Mean Difference (Net) = 28.833, 95% CI 2-sided [18.9550 to 38.7102] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 4: Comparison: Atorvastatin 10 mg + Ezetimibe 10 mg vs Placebo; For HDLc; Test type: Superiority or Other; Mean Difference (Net) = 3.701, 95% CI 2-sided [-5.5562 to 12.9578] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 5: Comparison: Atorvastatin 80 mg + GSK1292263 800 mg vs Placebo; For HDLc; Test type: Superiority or Other; Mean Difference (Net) = 20.946, 95% CI 2-sided [8.6120 to 33.2810] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 6: Comparison: GSK1292263 100 mg vs Placebo; For HDLc; Test type: Superiority or Other; Median Difference (Net) = 10.561, 95% CI 2-sided [-0.9675 to 22.0898] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 7: Comparison: GSK1292263 300 mg vs Placebo; For HDLc; Test type: Superiority or Other; Mean Difference (Net) = 11.122, 95% CI 2-sided [-0.2902 to 22.5351] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 8: Comparison: GSK1292263 800 mg vs Placebo; For HDLc; Test type: Superiority or Other; Mean Difference (Net) = 20.689, 95% CI 2-sided [9.7527 to 31.6262] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 9: Comparison: Atorvastatin 10 mg + GSK1292263 100 mg vs Placebo; For LDLc; Test type: Superiority or Other; Mean Difference (Net) = -4.549, 95% CI 2-sided [-18.7750 to 9.6768] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 10: Comparison: Atorvastatin 10 mg + GSK1292263 300 mg vs Placebo; For LDLc; Test type: Superiority or Other; Mean Difference (Net) = -10.337, 95% CI 2-sided [-24.4549 to 3.7803] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 11: Comparison: Atorvastatin 10 mg + GSK1292263 800 mg vs Placebo; For LDLc; Test type: Superiority or Other; Mean Difference (Net) = -21.317, 95% CI 2-sided [-36.0144 to -6.6190] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 12: Comparison: Atorvastatin 10 mg + Ezetimibe 10 mg vs Placebo; For LDLc; Test type: Superiority or Other; Mean Difference (Net) = -20.173, 95% CI 2-sided [-34.2710 to -6.0755] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 13: Comparison: Atorvastatin 80 mg + GSK1292263 800 mg vs Placebo; For LDLc; Test type: Superiority or Other; Mean Difference (Net) = -25.472, 95% CI 2-sided [-49.3385 to -8.1558] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 14: Comparison: GSK1292263 100 mg vs Placebo; For LDLc; Test type: Superiority or Other; Mean Difference (Net) = -12.128, 95% CI 2-sided [-23.3049 to -0.9514] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 15: Comparison: GSK1292263 300 mg vs Placebo; For LDLc; Test type: Superiority or Other; Mean Difference (Net) = -15.798, 95% CI 2-sided [-27.1364 to -4.4589] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 16: Comparison: GSK1292263 800 mg vs Placebo; For LDLc; Test type: Superiority or Other; Mean Difference (Net) = -21.789, 95% CI 2-sided [-32.3413 to -11.2372] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 17: Comparison: Atorvastatin 10 mg + GSK1292263 100 mg vs Placebo; For Triglycerides; Test type: Superiority or Other; Mean Difference (Net) = -22.498, 95% CI 2-sided [-38.4460 to -2.4169] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 18: Comparison: Atorvastatin 10 mg + GSK1292263 300 mg vs Placebo; For Triglycerides; Test type: Superiority or Other; Mean Difference (Net) = -23.781, 95% CI 2-sided [-39.1603 to -4.5130] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 19: Comparison: Atorvastatin 10 mg + GSK1292263 800 mg vs Placebo; For Triglycerides; Test type: Superiority or Other; Mean Difference (Net) = -39.923, 95% CI 2-sided [-52.3394 to -24.2717] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 20: Comparison: Atorvastatin 10 mg + Ezetimibe 10 mg vs Placebo; For Triglycerides; Test type: Superiority or Other; Mean Difference (Net) = -17.444, 95% CI 2-sided [-33.5020 to 2.4910] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 21: Comparison: Atorvastatin 80 mg + GSK1292263 800 mg vs Placebo; For Triglycerides; Test type: Superiority or Other; Mean Difference (Net) = -21.781, 95% CI 2-sided [-40.2960 to -3.2667] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 22: Comparison: GSK1292263 100 mg vs Placebo; For Triglycerides; Test type: Superiority or Other; Mean Difference (Net) = -21.421, 95% CI 2-sided [-38.3519 to -4.4911] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 23: Comparison: GSK1292263 300 mg vs Placebo; For Triglycerides; Test type: Superiority or Other; Mean Difference (Net) = -46.361, 95% CI 2-sided [-63.4650 to -29.2561] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 24: Comparison: GSK1292263 800 mg vs Placebo; For Triglycerides; Test type: Superiority or Other; Mean Difference (Net) = -54.843, 95% CI 2-sided [-70.7854 to -38.9007] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 25: Comparison: Atorvastatin 10 mg + GSK1292263 100 mg vs Placebo; For Non-HDLc; Test type: Superiority or Other; Mean Difference (Net) = -9.756, 95% CI 2-sided [-21.7561 to 2.2448] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 26: Comparison: Atorvastatin 10 mg + GSK1292263 300 mg vs Placebo; For Non-HDLc; Test type: Superiority or Other; Mean Difference (Net) = -14.014, 95% CI 2-sided [-25.7497 to -2.2787] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 27: Comparison: Atorvastatin 10 mg + GSK1292263 800 mg vs Placebo; For Non-HDLc; Test type: Superiority or Other; Mean Difference (Net) = -27.675, 95% CI 2-sided [-39.8454 to -15.5045] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 28: Comparison: Atorvastatin 10 mg + Ezetimibe 10 mg vs Placebo; For Non-HDLc; Test type: Superiority or Other; Mean Difference (Net) = -20.937, 95% CI 2-sided [-32.6057 to -9.2690] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 29: Comparison: Atorvastatin 80 mg + GSK1292263 800 mg vs Placebo; For Non-HDLc; Test type: Superiority or Other; Mean Difference (Net) = -21.702, 95% CI 2-sided [-29.0346 to -14.3696] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 30: Comparison: GSK1292263 100 mg vs Placebo; For Non-HDLc; Test type: Superiority or Other; Mean Difference (Net) = -13.180, 95% CI 2-sided [-23.0636 to -3.2961] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 31: Comparison: GSK1292263 300 mg vs Placebo; For Non-HDLc; Test type: Superiority or Other; Mean Difference (Net) = -22.151, 95% CI 2-sided [-31.9420 to -12.3605] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 32: Comparison: GSK1292263 800 mg vs Placebo; For Non-HDLc; Test type: Superiority or Other; Mean Difference (Net) = -26.948, 95% CI 2-sided [-36.2874 to -17.6092] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 33: Comparison: Atorvastatin 10 mg + GSK1292263 100 mg vs Placebo; For Cholesterol; Test type: Superiority or Other; Mean Difference (Net) = -3.904, 95% CI 2-sided [-11.8484 to 4.0400] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 34: Comparison: Atorvastatin 10 mg + GSK1292263 300 mg vs Placebo; For Cholesterol; Test type: Superiority or Other; Mean Difference (Net) = -6.437, 95% CI 2-sided [-14.3460 to 1.4722] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 35: Comparison: Atorvastatin 10 mg + GSK1292263 800 mg vs Placebo; For Cholesterol; Test type: Superiority or Other; Mean Difference (Net) = -10.294, 95% CI 2-sided [-18.3923 to -2.1960] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 36: Comparison: Atorvastatin 10 mg + Ezetimibe 10 mg vs Placebo; For Cholesterol; Test type: Superiority or Other; Mean Difference (Net) = -12.065, 95% CI 2-sided [-19.7688 to -4.3609] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 37: Comparison: Atorvastatin 80 mg + GSK1292263 800 mg vs Placebo; For Cholesterol; Test type: Superiority or Other; Mean Difference (Net) = -7.941, 95% CI 2-sided [-13.9778 to -1.9039] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 38: Comparison: GSK1292263 100 mg vs Placebo; For Cholesterol; Test type: Superiority or Other; Mean Difference (Net) = -8.384, 95% CI 2-sided [-15.9023 to -0.8660] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 39: Comparison: GSK1292263 300 mg vs Placebo; For Cholesterol; Test type: Superiority or Other; Mean Difference (Net) = -15.700, 95% CI 2-sided [-23.1404 to -8.2592] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 40: Comparison: GSK1292263 800 mg vs Placebo; For Cholesterol; Test type: Superiority or Other; Mean Difference (Net) = -16.728, 95% CI 2-sided [-23.8395 to -9.6161]

40. Primary Outcome: Percent Change From Baseline in Lipid Metabolism: LDL/HDL Ratio at Day 14 (24 Hours)
Description: as for outcome 37
Time Frame: Baseline and Day 14
Population: All subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo | GSK1292263 100 mg | GSK1292263 300 mg | GSK1292263 800 mg | Placebo
Number analyzed (Participants) | 11 | 11 | 10 | 12 | 13 | 11 | 12 | 10 | 11 | 13 | 10
Percent change | -12.25 (14.784) | -21.12 (20.549) | -41.61 (14.248) | 0.94 (20.727) | -28.69 (11.963) | -34.35 (16.047) | 10.84 (56.487) | -16.78 (15.615) | -17.63 (23.327) | -32.01 (11.287) | 2.55 (12.789)
Statistical Analysis 1: Comparison: Atorvastatin 10 mg + GSK1292263 100 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -12.123, 95% CI 2-sided [-26.6276 to 2.3814] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 2: Comparison: Atorvastatin 10 mg + GSK1292263 300 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -21.630, 95% CI 2-sided [-35.9419 to -7.3181] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 3: Comparison: Atorvastatin 10 mg + GSK1292263 800 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -41.506, 95% CI 2-sided [-56.3924 to -26.6205] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 4: Comparison: Atorvastatin 10 mg + Ezetimibe 10 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -28.041, 95% CI 2-sided [-42.2554 to -13.8263] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 5: Comparison: Atorvastatin 80 mg + GSK1292263 800 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -29.293, 95% CI 2-sided [-51.5654 to -12.4042] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 6: Comparison: GSK1292263 100 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -20.042, 95% CI 2-sided [-34.8358 to -5.2472] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 7: Comparison: GSK1292263 300 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -21.903, 95% CI 2-sided [-36.6155 to -7.1913] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 8: Comparison: GSK1292263 800 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -35.735, 95% CI 2-sided [-49.7220 to -21.7485] — Statistical analysis was performed using LS mean value of GSK1292263

41. Primary Outcome: Weighted Mean Area Under Concentration Curve From 0 to 24 Hours (AUC [0-24]) Change From Baseline for Triglycerides at Day 14
Description: Blood samples were collected fasting on Days 1 (pre-dose), 7 and 15 prior to checkout (24 hours post-dose), and at Follow-up. When this results in multiple samples at the same time point, only one sample will be collected (example, when 24 hours post-dose = pre-dose (time 0) for the next dose). Baseline was Day -1 value. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. If either the Baseline or post-randomization value is missing, the change from Baseline was set to missing as well. Percent change from Baseline was calculated as the change from Baseline divided by the Baseline value then multiplied by 100.
Time Frame: Baseline and Day 14
Population: All subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: millimoles per liter
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo | GSK1292263 100 mg | GSK1292263 300 mg | GSK1292263 800 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 12 | 13 | 11 | 13 | 10 | 12 | 13 | 11
millimoles per liter | 0.13341 (-167.395) | 0.30812 (-360.966) | 0.12845 (-68.4294) | 0.25228 (477.0380) | 0.09060 (-146.956) | 0.04974 (-76.1973) | 0.20164 (-485.961) | 0.30543 (-159.012) | 0.37442 (-111.818) | 0.13079 (-115.210) | 0.28863 (93.3050)
Statistical Analysis 1: Comparison: Atorvastatin 10 mg + GSK1292263 100 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.409, 95% CI 2-sided [-1.0123 to 0.1942] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 2: Comparison: Atorvastatin 10 mg + GSK1292263 300 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.296, 95% CI 2-sided [-0.9063 to 0.3141] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 3: Comparison: Atorvastatin 10 mg + GSK1292263 800 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.811, 95% CI 2-sided [-1.4125 to -0.2098] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 4: Comparison: Atorvastatin 10 mg + Ezetimibe 10 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.422, 95% CI 2-sided [-0.9831 to 0.1394] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 5: Comparison: Atorvastatin 80 mg + GSK1292263 800 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.384, 95% CI 2-sided [-0.6009 to -0.1669] — Statistical analysis was performed using LS mean value of Atorvastatin
Statistical Analysis 6: Comparison: GSK1292263 100 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.648, 95% CI 2-sided [-1.1657 to -0.1302] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 7: Comparison: GSK1292263 300 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.782, 95% CI 2-sided [-1.2804 to -0.2844] — Statistical analysis was performed using LS mean value of GSK1292263
Statistical Analysis 8: Comparison: GSK1292263 800 mg vs Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.884, 95% CI 2-sided [-1.3652 to -0.4026] — Statistical analysis was performed using LS mean value of GSK1292263

42. Secondary Outcome: Cmax of Atorvastatin Metabolite (2-Hydroxyatorvastatin)- Part A
Description: Serial blood samples for the determination of the PK for atorvastatin metabolites on Day -1 was collected at immediately pre-morning dose=pre-breakfast (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14 and 24 hours post-morning dose (24 hour sample Day -1 = 0 hour sample Day 1). Serial blood samples for the determination of the PK for atorvastatin metabolites on Days 1 and 14 will be collected at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hour post-morning dose (no 48h sample on Day 1).
Time Frame: as for outcome 30
Population: PK parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Atorvastatin 80 mg + GSK1292263 800 mg
Number analyzed (Participants) | 4
nanograms per milliliter
  Day -1 | 17.521 (66.1066)
  Day 1 | 15.535 (48.2576)
  Day 14 | 21.271 (30.4382)

43. Secondary Outcome: Cmax of Atorvastatin Metabolite (2-Hydroxyatorvastatin)- Part B (Pooled Treatment Arm)
Description: For co-dosing arms, serial blood samples for the determination of the PK of atorvastatin metabolites were collected on Day -1 and for atorvastatin metabolites on Days 1 and 14. Blood samples for PK were collected on Days -1 (co-dosing arms only) and 1 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, and 24 hours post-morning dose. Blood samples for PK were collected on Day 14 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hours post-morning dose (48 hour PK sample was collected on Day 16).
Time Frame: as for outcome 31
Population: PK parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo
Number analyzed (Participants) | 7 | 7 | 11 | 12 | 6 | 12 | 13
nanograms per milliliter
  Day -1: number analyzed (Participants) | 4 | 5 | 10 | 12 | 6 | 12 | 13
  Day -1 | 1.298 (37.3615) | 1.388 (42.8163) | 0.947 (39.3947) | 0.952 (63.1814) | 1.185 (119.9675) | 26.106 (102.2617) | 21.149 (39.5618)
  Day 1: number analyzed (Participants) | 4 | 5 | 11 | 12 | 5 | 12 | 13
  Day 1 | 1.073 (19.3329) | 1.217 (36.0597) | 1.048 (33.9165) | 1.028 (67.0630) | 1.234 (44.7679) | 19.991 (71.2442) | 26.400 (44.9589)
  Day 14: number analyzed (Participants) | 4 | 5 | 10 | 12 | 5 | 11 | 13
  Day 14 | 0.634 (12.5545) | 1.152 (53.4256) | 1.084 (49.9097) | 0.869 (62.0112) | 1.349 (42.0203) | 22.645 (75.7161) | 27.236 (68.7891)

44. Secondary Outcome: Tmax of Atorvastatin Metabolite (2-Hydroxyatorvastatin)- Part A
Description: as for outcome 42
Time Frame: as for outcome 30
Population: PK parameter Population.
Measure: Median (Full Range); unit: hours
Arm/Group | Atorvastatin 80 mg + GSK1292263 800 mg
Number analyzed (Participants) | 4
hours
  Day -1 | 3.000 [1.00 to 4.00]
  Day 1 | 4.000 [4.00 to 6.00]
  Day 14 | 2.500 [2.00 to 4.00]

45. Secondary Outcome: Tmax of Atorvastatin Metabolite (2-Hydroxyatorvastatin)- Part B (Pooled Treatment Arm)
Description: as for outcome 43
Time Frame: On Days -1 and 1 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, and 24 hours post-morning dose and on Day 14 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hours post-morning dose
Population: PK parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo
Number analyzed (Participants) | 7 | 7 | 11 | 12 | 6 | 12 | 13
hours
  Day -1: number analyzed (Participants) | 4 | 5 | 10 | 12 | 6 | 12 | 13
  Day -1 | 4.500 [1.00 to 6.08] | 4.000 [3.00 to 8.00] | 5.000 [2.00 to 8.02] | 4.000 [3.00 to 8.00] | 4.000 [4.00 to 6.00] | 3.992 [1.00 to 6.00] | 3.000 [1.00 to 4.00]
  Day 1: number analyzed (Participants) | 4 | 5 | 11 | 12 | 5 | 12 | 13
  Day 1 | 6.000 [6.00 to 6.00] | 6.000 [4.00 to 8.00] | 4.000 [2.00 to 14.10] | 4.000 [1.50 to 10.00] | 4.000 [2.00 to 6.00] | 4.000 [1.50 to 6.08] | 3.000 [0.50 to 6.02]
  Day 14: number analyzed (Participants) | 4 | 5 | 10 | 12 | 5 | 11 | 13
  Day 14 | 6.000 [2.83 to 8.00] | 4.000 [3.00 to 14.00] | 4.025 [3.00 to 6.08] | 5.000 [1.50 to 14.02] | 6.000 [3.00 to 6.00] | 4.000 [1.50 to 6.00] | 3.983 [1.00 to 6.05]

46. Secondary Outcome: AUC (0-24) of Atorvastatin Metabolite (2-Hydroxyatorvastatin)- Part A
Description: as for outcome 42
Time Frame: as for outcome 30
Population: PK parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms hour per milliliter
Arm/Group | Atorvastatin 80 mg + GSK1292263 800 mg
Number analyzed (Participants) | 4
nanograms hour per milliliter
  Day -1 | 119.66 (72.635)
  Day 1 | 127.70 (49.098)
  Day 14 | 139.78 (47.491)

47. Secondary Outcome: AUC (0-24) of Atorvastatin Metabolite (2-Hydroxyatorvastatin)- Part B (Pooled Treatment Arm)
Description: as for outcome 43
Time Frame: as for outcome 31
Population: PK parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms hour per milliliter
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo
Number analyzed (Participants) | 7 | 7 | 11 | 12 | 6 | 12 | 13
nanograms hour per milliliter
  Day -1: number analyzed (Participants) | 3 | 5 | 9 | 11 | 6 | 11 | 12
  Day -1 | 16.72 (19.509) | 20.25 (47.047) | 14.37 (48.598) | 12.38 (74.286) | 12.41 (53.128) | 163.16 (73.666) | 133.96 (36.159)
  Day 1: number analyzed (Participants) | 4 | 5 | 11 | 11 | 5 | 11 | 13
  Day 1 | 16.02 (9.355) | 18.28 (40.611) | 14.89 (33.541) | 13.60 (78.379) | 15.10 (26.181) | 146.23 (55.353) | 150.41 (37.440)
  Day 14: number analyzed (Participants) | 3 | 5 | 9 | 12 | 4 | 11 | 13
  Day 14 | 10.07 (12.346) | 16.54 (37.123) | 13.82 (43.131) | 12.03 (63.145) | 18.18 (36.758) | 144.23 (58.954) | 156.41 (42.286)

48. Secondary Outcome: Trough Concentration of Atorvastatin Metabolite (2-Hydroxyatorvastatin)
Description: For co-dosing arms, serial blood samples for the determination of the PK of atorvastatin metabolites were supposed to collected on Day -1 and for atorvastatin metabolites on Days 1 and 14. Blood samples for PK were supposed to collected on Days -1 (co-dosing arms only) and 1 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, and 24 hours post-morning dose. Blood samples for PK were supposed to collected on Day 14 at immediately pre-morning dose (time 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 14, 24 and 48 hours post-morning dose (48 hour PK sample was collected on Day 16). However no data was collected.
Time Frame: as for outcome 31
Arm/Group | Atorvastatin 10 mg + GSK1292263 100 mg | Atorvastatin 10 mg + GSK1292263 300 mg | Atorvastatin 10 mg + GSK1292263 800 mg | Atorvastatin 10 mg + Placebo | Atorvastatin 10 mg + Ezetimibe 10 mg | Atorvastatin 80 mg + GSK1292263 800 mg | Atorvastatin 80 mg + Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All AEs and SAEs were collected up to follow-up visit. For Part A- up to Day 26, for Part B (washout)- up to Day 28, for Part B (run-in)- up to day up to day 28 and Part B (treatment)- up to Day 26
Description: All AEs and SAEs for Part A were collected using Safety Population and for Part B using All Subjects Population.
Groups:
- 80 mg Atorvastatin + 800 mg GSK1292263 (Part A): Participants on 80 mg atorvastatin (either for >=4 weeks prior to screening (80 mg), or for 2 weeks, if the dose was escalated from a stable dose of 40 mg) received 800 mg of GSK1292263 for 2 weeks once daily immediately after eating the breakfast meal.
- 800 mg GSK1292263 (Part A): Participants not on lipid-modifying treatment received GSK1282263 alone for 2 weeks once daily immediately after eating the breakfast meal.
- Pre-treatment (Part B): This was the time period prior to Day 1 of Washout Phase.
- Washout (Part B): During the 4 weeks washout period, participants were asked to stop their lipid-modifying drugs.
- Atorvastatin 10 mg (Part B Run-in): After washout participants received atorvastatin 10 mg for a 4-week stabilization Run-in Period.
- Atorvastatin 80 mg (Part B Run-in): After washout participants received atorvastatin 80 mg for a 4-week stabilization Run-in Period.
- Atorvastatin 10 mg + GSK1292263 100 mg (Part B Treatment): Participants received 10 mg atorvastatin along with GSK1292263 100 mg once daily for 2 weeks.
- Atorvastatin 10 mg + GSK1292263 300 mg (Part B Treatment): Participants received 10 mg atorvastatin along with GSK1292263 300 mg once daily for 2 weeks.
- Atorvastatin 10 mg + GSK1292263 800 mg (Part B Treatment): Participants received 10 mg atorvastatin along with GSK1292263 800 mg once daily for 2 weeks.
- Atorvastatin 10 mg + Placebo (Part B Treatment): Participants received 10 mg atorvastatin along with placebo matching to GSK1292263 once daily for 2 weeks.
- Atorvastatin 10 mg + Ezetimibe 10 mg (Part B Treatment): Participants received 10 mg atorvastatin along with Ezetimibe 10 mg once daily for 2 weeks.
- Atorvastatin 80 mg + GSK1292263 800 mg (Part B Treatment): Participants received 80 mg atorvastatin along with GSK1292263 800 mg once daily for 2 weeks.
- Atorvastatin 80 mg + Placebo (Part B Treatment): Participants received 80 mg atorvastatin along with placebo matching to GSK1292263 once daily for 2 weeks.
- GSK1292263 100 mg (Part B Treatment): After washout, participants were randomized to receive monotherapy of GSK1292263 100 mg once daily for 2 weeks.
- GSK1292263 300 mg (Part B Treatment): After washout, participants were randomized to receive monotherapy of GSK1292263 300 mg once daily for 2 weeks.
- GSK1292263 800 mg (Part B Treatment): After washout, participants were randomized to receive monotherapy of GSK1292263 800 mg once daily for 2 weeks.
- Placebo (Part B Treatment): After washout, participants were randomized to receive placebo matching to GSK1292263 once daily for 2 weeks.
Arm/Group | 80 mg Atorvastatin + 800 mg GSK1292263 (Part A) | 800 mg GSK1292263 (Part A) | Pre-treatment (Part B) | Washout (Part B) | Atorvastatin 10 mg (Part B Run-in) | Atorvastatin 80 mg (Part B Run-in) | Atorvastatin 10 mg + GSK1292263 100 mg (Part B Treatment) | Atorvastatin 10 mg + GSK1292263 300 mg (Part B Treatment) | Atorvastatin 10 mg + GSK1292263 800 mg (Part B Treatment) | Atorvastatin 10 mg + Placebo (Part B Treatment) | Atorvastatin 10 mg + Ezetimibe 10 mg (Part B Treatment) | Atorvastatin 80 mg + GSK1292263 800 mg (Part B Treatment) | Atorvastatin 80 mg + Placebo (Part B Treatment) | GSK1292263 100 mg (Part B Treatment) | GSK1292263 300 mg (Part B Treatment) | GSK1292263 800 mg (Part B Treatment) | Placebo (Part B Treatment)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2 | 0/281 | 0/281 | 0/62 | 0/27 | 0/11 | 0/11 | 0/11 | 0/12 | 0/13 | 0/12 | 0/13 | 0/11 | 0/12 | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 0/281 | 0/281 | 0/62 | 0/27 | 0/11 | 0/11 | 0/11 | 0/12 | 0/13 | 0/12 | 0/13 | 0/11 | 0/12 | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 0/4 | 2/2 | 14/281 | 37/281 | 19/62 | 8/27 | 6/11 | 2/11 | 3/11 | 3/12 | 4/13 | 6/12 | 4/13 | 5/11 | 7/12 | 8/13 | 4/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 80 mg Atorvastatin + 800 mg GSK1292263 (Part A) (N=4) | 800 mg GSK1292263 (Part A) (N=2) | Pre-treatment (Part B) (N=281) | Washout (Part B) (N=281) | Atorvastatin 10 mg (Part B Run-in) (N=62) | Atorvastatin 80 mg (Part B Run-in) (N=27) | Atorvastatin 10 mg + GSK1292263 100 mg (Part B Treatment) (N=11) | Atorvastatin 10 mg + GSK1292263 300 mg (Part B Treatment) (N=11) | Atorvastatin 10 mg + GSK1292263 800 mg (Part B Treatment) (N=11) | Atorvastatin 10 mg + Placebo (Part B Treatment) (N=12) | Atorvastatin 10 mg + Ezetimibe 10 mg (Part B Treatment) (N=13) | Atorvastatin 80 mg + GSK1292263 800 mg (Part B Treatment) (N=12) | Atorvastatin 80 mg + Placebo (Part B Treatment) (N=13) | GSK1292263 100 mg (Part B Treatment) (N=11) | GSK1292263 300 mg (Part B Treatment) (N=12) | GSK1292263 800 mg (Part B Treatment) (N=13) | Placebo (Part B Treatment) (N=11)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 5 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 7 | 7 | 1 | 3 | 1 | 1 | 0 | 2 | 2 | 3 | 2 | 1 | 2 | 2
Migraine (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.